CLINICAL TRIAL: NCT04505553
Title: Pilot Study of Oral Cryotherapy vs. Oral Cryotherapy Plus Acupuncture and Acupressure to Decrease Chemotherapy-Induced Peripheral Neuropathy From Oxaliplatin-Based Chemotherapy for GI Cancers
Brief Title: Oral Cryotherapy Plus Acupressure and Acupuncture Versus Oral Cryotherapy for Decreasing Chemotherapy-Induced Peripheral Neuropathy From Oxaliplatin-Based Chemotherapy in Patients With Gastrointestinal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Safeway Foundation (Unknown)
Responsible Party: Principal Investigator, Stacey Cohen, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1121095; NCI-2020-05455 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); 10559 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Appendix Carcinoma; Colon Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Liver and Intrahepatic Bile Duct Carcinoma; Malignant Digestive System Neoplasm; Pancreatic Carcinoma; Rectal Carcinoma; Small Intestinal Carcinoma; Anal Carcinoma; Digestive System Carcinoma; Digestive System Neuroendocrine Tumor; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Appendiceal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Gastro-enteropancreatic neuroendocrine tumor; Adenoma, Islet Cell | interventions — Acupuncture Therapy; Acupressure; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (acupuncture, acupressure, cryotherapy) (Experimental): Patients undergo acupuncture during chemotherapy infusion on day 1 and fluorouracil pump disconnect on day 3 of each biweekly chemotherapy infusion over 12 weeks. Patients also undergo self-administered acupressure over 11 minutes daily for 12 weeks and undergo standard of care oral cryotherapy.
  Interventions: Procedure: Acupuncture Therapy; Procedure: Acupressure Therapy; Procedure: Oral Cryotherapy; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (cryotherapy) (Active Comparator): Patients undergo standard of care oral cryotherapy.
  Interventions: Procedure: Oral Cryotherapy; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Acupuncture Therapy — Undergo acupuncture
  Other Names: Acupuncture
  Arms: Arm I (acupuncture, acupressure, cryotherapy)
Procedure: Acupressure Therapy — Undergo acupressure
  Other Names: acupressure; Ischemic Compression
  Arms: Arm I (acupuncture, acupressure, cryotherapy)
Procedure: Oral Cryotherapy — Undergo oral cryotherapy
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial investigates how well oral cryotherapy plus acupressure and acupuncture compared with oral cryotherapy alone work in decreasing chemotherapy-induced peripheral neuropathy in patients with gastrointestinal cancer who are receiving oxaliplatin-based chemotherapy. Acupressure is the application of pressure or localized massage to specific sites on the body to control symptoms such as pain or nausea. Acupuncture is the technique of inserting thin needles through the skin at specific points on the body to control pain and other symptoms. Cryotherapy uses cold temperature such as oral ice chips to prevent abnormally increased pain sensation. Giving oral cryotherapy with acupressure and acupuncture may work better in decreasing chemotherapy-induced peripheral neuropathy from oxaliplatin-based chemotherapy in patients with gastrointestinal cancer compared to oral cryotherapy alone.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo acupuncture during chemotherapy infusion on day 1 and fluorouracil pump disconnect on day 3 of each biweekly chemotherapy infusion over 12 weeks. Patients also undergo self-administered acupressure over 11 minutes daily for 12 weeks and undergo standard of care oral cryotherapy.

ARM II: Patients undergo standard of care oral cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* GI cancer (primary esophagus, gastric, pancreas, biliary, liver, small bowel, appendix, colon, rectal, anal, or gastrointestinal/pancreatic neuroendocrine tumor) scheduled to receive a new start of fluorouracil (5-FU), oxaliplatin, +/- irinotecan (fluorouracil/leucovorin calcium/oxaliplatin [FOLFOX], fluorouracil/irinotecan/leucovorin calcium/oxaliplatin [FOLFIRINOX], leucovorin/fluorouracil/oxaliplatin/irinotecan [FOLFOXIRI] regimens) with plan for >= 3 months of therapy with the regimen. Chemotherapy can be given for neoadjuvant, adjuvant, or palliative intent. 1 dose (cycle) of the intended regimen is permitted prior to study enrollment.

  **There is no limitation on the addition of a biologic agent to one of the above chemotherapy regimens, including, but not limited to: bevacizumab, cetuximab, panitumumab, trastuzumab, or the biosimilars of these agents
* Age >=18 years
* Absolute neutrophil count > 0.5 thousand/microL
* Platelet count > 20 thousand/microL
* Not currently pregnant
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Baseline peripheral neuropathy from any cause
* Planned oxaliplatin with capecitabine
* Planned initial dose of oxaliplatin < 100% of the standard regimen-specified dose. For most regimens, this would be 85 mg/m^2 intravenously (IV) dosed every 14 days
* Receipt of acupuncture treatment in the prior 3 months
* Use of concomitant duloxetine for minimization of neuropathy
* Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Cohen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Started | 37 | 41
Completed | 33 | 36
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy) | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 36 | 68
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 24 | 26 | 50
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 36 | 69
European Organisation For Research & Treatment of Cancer-CIPN 20 questionnaire [Mean (Standard Deviation); unit: units on a scale] — EORTC (European Organisation For Research And Treatment Of Cancer) CIPN (Chemotherapy-Induced Peripheral Neuropathy) 20 QOL (Quality of Life Questionnaire) patient reported outcomes questionnaire was used. 3 subscales all scored from 1 to 4: Sensory, Motor, and Autonomic. For all subscales: higher values represent a worse outcome. All subscales are to be reported separately. The raw scores are linearly converted to a 0-100 scale such that a higher score corresponds to a worse condition or more symptoms.
  units on a scale
    Sensory | 35 (3.7) | 36.4 (4.5) | 35.8 (4.2)
    Motor | 36.5 (5.9) | 36.8 (6.6) | 36.6 (6.2)
    Autonomic | 37.8 (11.6) | 45.3 (16.7) | 42.1 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Chemotherapy-induced Peripheral Neuropathy (CIPN) From Baseline to 3 Months
Description: Measured by the European Organization for Research and Treatment of Cancer (EORTC)-CIPN 20. Severity of CIPN will be summarized for each treatment arm, and treatment comparisons made via linear regression model with adjustment for baseline severity level. The EORTC QLQ-CIPN20 is a 20-item questionnaire that evaluates CIPN using 3 subscales that assess sensory (9 items), motor (8 items), and autonomic (3 items) symptoms and functioning. The CIPN-20 subscale raw scores are linearly converted to a 0-100 scale such that a high score corresponds to a worse condition or more symptoms. Change in severity was measured by the difference in the converted scores from baseline to three months and the range is -100 to 100.
Time Frame: At 3 months
Population: Due to missing patient reported outcomes the overall number of participants analyzed differs from patients that completed the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Number analyzed (Participants) | 20 | 27
units on a scale
  Sensory Subscale | 5.9 [-7.4 to 37.0] | 9.1 [-11.1 to 25.9]
  Motor Subscale | 1.9 [-16.7 to 12.5] | 5.7 [-4.2 to 25.0]
  Autonomic Subscale | 0.6 [-33.3 to 22.2] | 0.8 [-50.0 to 44.4]

2. Secondary Outcome: Number of Participants With Grade 2 or Higher Chemotherapy-Induced Peripheral Neuropathy
Description: Measured by Common Terminology Criteria for Adverse Events (CTCAE) version 5. Incidences of CIPN (grade 2 or higher), pain, fatigue, nausea, and anxiety will be compared between treatment arms using Chi-squared or Fisher's exact tests as appropriate.
Time Frame: 3 months
Population: Frequency of Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Number analyzed (Participants) | 33 | 36
Participants
  No Peripheral Sensory Neuropathy | 28 | 33
  Peripheral Sensory Neuropathy | 5 | 3

3. Secondary Outcome: Severity of CIPN: Neuropen Assessment of Patients' Perceived Pressure
Description: The Neuropen is used to assess pressure perception. Pressure sensation will be assessed using a 10-g monofilament on the subject's dominant foot at each of the ten different sites recorded as present or absent. The proportion present was calculated for each patient at baseline and at 3 months. The difference between these proportions from baseline to 3 months was calculated for each patient. The mean of these differences was calculated within each arm and the difference of those means was then compared between arms.
Time Frame: 3 months
Population: Due to missing acupuncture appointments the overall number of participants analyzed differs from patients that completed the study.
Measure: Mean (Standard Deviation); unit: proportion of present responses
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Number analyzed (Participants) | 21 | 27
proportion of present responses | -1.0 (4.4) | -0.7 (7.3)

4. Secondary Outcome: Severity of CIPN: Tuning Fork Vibration Sensation Testing
Description: A study-specific 128-Hz tuning fork will be used to assess vibration sensation on the great toe at baseline and 3 months. The time in seconds to loss of vibration sensation was measured. Vibration sensation is lost sooner in CIPN, which means that shorter duration of vibration scores are associated with increased CIPN. The difference from baseline to 3 months in number of seconds to loss of vibration sensation was calculated for each patient. The differences were averaged across patients in each arm. The mean differences were compared between arms.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Number analyzed (Participants) | 21 | 27
seconds | -5.0 (11.6) | 0.1 (6.6)

5. Secondary Outcome: Proportion of Patients Assigned to the Intervention Arm Who Complete 60% of Acupuncture Treatments
Description: Adherence to acupuncture treatment among patients in the intervention arm will be described as a proportion with 95% confidence interval. Reasons for treatment non-adherence and delivered dose intensity of chemotherapy will be noted.
Time Frame: 3 months
Population: Summary of Patient Adherence to Acupuncture Protocol Based on 60% Threshold
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy)
Number analyzed (Participants) | 33
Participants
  Adherent | 23
  Nonadherent | 10

6. Secondary Outcome: Change in Severity of Pain, Fatigue, Nausea, and Anxiety From Baseline to 3 Months
Description: Measured by patient-reported National Cancer Institute [NCI] Patient Reported Outcomes [PRO]-CTCAE. The change in severity from baseline to 3 months was calculated and it ranged from -3 to 3. The severity was measured on a 0-3 (0=None, 3=Severe) scale with a higher value representing a worse outcome and a lower value representing a better outcome. This was done separately for pain, fatigue, nausea, and anxiety.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
Number analyzed (Participants) | 20 | 27
units on a scale
  Pain: number analyzed (Participants) | 19 | 27
  Pain | -0.3 (1.2) | -0.3 (1.1)
  Fatigue | -0.1 (0.9) | 0.4 (1.2)
  Nausea: number analyzed (Participants) | 19 | 27
  Nausea | -0.3 (0.7) | 0.3 (1.0)
  Anxiety: number analyzed (Participants) | 19 | 27
  Anxiety | -0.1 (1.0) | -0.1 (0.9)

ADVERSE EVENTS:
Time Frame: 22 weeks
Description: CTCAE vr. 5 terms used
Arm/Group | Arm I (Acupuncture, Acupressure, Cryotherapy) | Arm II (Cryotherapy)
All-Cause Mortality (participants affected / at risk) | 5/33 | 3/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 18/33 | 26/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Acupuncture, Acupressure, Cryotherapy) (N=33) | Arm II (Cryotherapy) (N=36)
Nausea (Gastrointestinal disorders) | 17 | 22
Fatigue (General disorders) | 15 | 26
Anxiety (Psychiatric disorders) | 2 | 0
Oral Symptoms (Gastrointestinal disorders) | 7 | 8 — Reported as Dry mouth; Mucositis oral; Oral pain; or Oral dysesthesia
Abdominal Pain (Gastrointestinal disorders) | 5 | 10 — Reported as Abdominal pain and Dyspepsia
Other Body Pain (Musculoskeletal and connective tissue disorders) | 1 | 7 — 1 or more Events reported as Back pain, Muscle cramp, Pain in extremity, Non-cardiac chest pain
Dysgeusia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 1 | 8
Blurred Vision (Eye disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 14 | 13
Diarrhea (Gastrointestinal disorders) | 8 | 16
Dizziness (Nervous system disorders) | 0 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Edema Limbs (General disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Eye Pain (Eye disorders) | 0 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hot Flashes (Vascular disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Paresthesia (Nervous system disorders) | 7 | 12
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 18 | 20
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Other Surgical and Medical Procedures (Surgical and medical procedures) | 0 | 2 — Any surgery or procedure completed
Vomiting (Gastrointestinal disorders) | 8 | 9
Confusion (Psychiatric disorders) | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Neutrophil Count Decreased (Investigations) | 2 | 0
Platelet Count Decreased (Investigations) | 2 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 3 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
White Blood Cell Decreased (Investigations) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT04505553/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT04505553/ICF_000.pdf